CLINICAL TRIAL: NCT05292326
Title: Assessment of Safety and Efficiency of the Medical Device Called PacePress to Prevent Hemorrhagic Complications in Patients With High Bleeding Risk Undergoing CIED Implantation Procedures in an Open-label, Multi-Centre Clinical Trial.
Brief Title: Safety and Efficiency of the PacePress to Prevent Hemorrhagic Complications in Patients Undergoing CIED Implantation.
Acronym: PacePress
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped at interim analysis due to significantly better outcomes with PacePress, consistent with the predefined statistical methodology.
Sponsor: Medinice S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PacePress_2020_03
Record Dates: First submitted 2021-09-30; First posted 2022-03-23 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hemorrhagic Complications; Hematoma; Hemorrhage; Pathologic Processes
Keywords: CIED Implantation; Hemorrhagic Complications; hematoma; pocket hematoma; bleeding risk score; cardiac implantable electronic device
MeSH Terms: conditions — Hematoma; Hemorrhage; Pathologic Processes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PacePress (Experimental): the patients will be dressed with PacePress medical device instead of a standard compression device
  Interventions: Device: PacePress
- standard compression band/tourniquet (Active Comparator): standard treatment with respect to preventing hemorrhagic complications and implantation site inflammation, the patients will be dressed with a standard compression device/sand bag
  Interventions: Device: standard compression band

INTERVENTIONS:
Device: PacePress — an electronically-controlled compression site which, thanks to a well-selected compression force, may contribute significantly to preventing hemorrhagic complications following electrotherapy procedures, including to increasing safety of CIED implantation procedures and accelerate wound healing significantly
  Arms: PacePress
Device: standard compression band — standard used compression band/sand bag
  Arms: standard compression band/tourniquet

SUMMARY:
PacePress medical device, by ensuring constant compression force and the ability to optimize it in the pocket area prevents/significantly reduces the risk of hemorrhagic complications, including but not limited to the operation pocket hematoma. By avoiding a strong localized compression and ensuring "covering compression" achieved by the appropriate distribution of compression forces on the entire implantation site area, with an automated compression force control, the risk of a pressure sore created in the compressed pocket area is reduced.

DETAILED DESCRIPTION:
The study will be an open-label, multi-center, monitored randomized study with 235 subjects qualified for:

* the CIED implantation procedure (initial),
* the CIED replacement procedure (ICD, CRT),
* expantion of the system,
* revision of electrodes.

The study consists in randomization of patients who meet all the inclusion criteria and do not meet any of the exclusion criteria, after performing the above procedure for the group (A): the PacePress medical device will be used, or (B): a standard of care will be used, in order to compare the safety and efficacy of the PacePress in relation to the standard of care, in preventing hemorrhagic complications and site infections.

Data regarding the assessment of the safety and effectiveness of the PacePress medical device are collected on the day of the procedure and during the 30-day patient observation.

In PacePress clinical trial, the standard pharmacotherapeutic procedures in the facility are not modified or affected (including but not limited to the anti-coagulation and antiplatelet treatment) according to the guidelines and standard procedure ESC and PTK in patients included in the study.

The investigational medical device is the PacePress (Medinice S.A.). This is an electronically-controlled self-pressure dressing that, , thanks to a well-selected compression force, may contribute significantly to preventing hemorrhagic complications following electrotherapy procedures, including increasing the safety of CIED implantation procedures and accelerating wound healing significantly.

The planned number of patients included in the study is 235 patients aged above 18 years. The study subjects will be divided into groups at random (4:1):

GROUP A - Following the procedure, the patients will be dressed in the PacePress - investigational medical device instead of a standard compression device.

The planned number of group members: n= 188 people.

GROUP B - Following the procedure, the patients will be dressed in the standard compression device.

The planned number of group members: n= 47 people.

In the study, the assumptions were made concerning the gradation and frequency of hematoma occurrence in particular groups and randomization of patients (4:1). Assuming the first-type error α=0.025 for the one-sided hypothesis and the test power of 0.8, 194 patients should be included in the study. Due to the planned interim analysis, which will be performed after half of the patients have been included in the study, and assuming the drop-out rate of 8 %, the required sample size should be increased to 235 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. The patient qualified for:

   * the CIED implantation procedure (initial),
   * the CIED replacement procedure (ICD, CRT),
   * expansion of the system,
   * revision of electrodes.
3. The patient standing high bleeding risk defined as a result of PACE DRAP ≥5.
4. The patient taking anti-coagulation or anti-platelet drugs or anti-coagulation and anti-platelet drugs permanently.

Exclusion Criteria:

1. The absence of written consent to participate in the study.
2. A female patient who is pregnant or breast-feeds.
3. The interview reveals addiction to alcohol, drugs, and other psychoactive substances.
4. The anamnesis reveals known hemorrhagic diathesis or thrombocytopenia, particularly after heparin is administered.
5. Active infection of the implantation site.
6. Active infection 4 weeks before inclusion in the study.
7. Anomaly in the chest near the device site.
8. The patient participates in another clinical trial.
9. Anticipated life span < 6 months.
10. Diagnosed allergy to any device ingredient.
11. The patient undergoes active biological therapy.
12. Treated cancer.
13. The patient undergoes shoulder girdle physiotherapy.
14. The patient undergoes systemic steroid therapy (intravenous therapy).
15. Obesity preventing the application of PacePress device.

    Criteria excluding the patient from the study that may appear during or immediately after the procedure:
16. Cardiac arrest (CPR)
17. Perforation.
18. Pneumothorax.
19. Intubation (patient intubated after the procedure).
20. Change of pacemaker position (conversion to the right side).
21. Procedure completed without implantation of the intended system.
22. Need for invasive treatment of complications of the procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Assessment of hematoma presence | 7 (-0/+2) days after the procedure
  according to the classification: Degree 0 - No hematoma Degree 1 - Hematoma not visible clinically - petechia above the device site (a tiny exudate or extravasation near the device, not causing any skin raising visible in a macroscopic scale), Degree 2 - Hematoma visible clinically - a visible macroscopically and palpable swelling of CIED area clearly exceeding the device dimensions, causing the tenderness and painfulness of the affected area; petechia going beyond the pocket, fluctuation symptom, small skin tension, small skin raising, Degree 3 - Hematoma significant clinically - much exceeding the device dimensions, causing significant skin tension and raising, requiring evacuation or extending hospital stay by at least 24 hours; pocket pain, significant skin raising.

SECONDARY OUTCOMES:
Emergence of a hematoma | based on 24-48 hour and 30 (+/- 5) day observation
  requiring a revision
Emergence of a hematoma | based on 24-48 hour, 7 (-0/+2) day and 30 (+/- 5) day observation
  requiring longer hospital stay
Number of patients who need blood derivative transfusion | based on 24-48 hour, 7 (-0/+2) day and 30 (+/- 5) day observation
  blood derivative transfusion need
Mortality rate | based on 24-48 hour, 7 (-0/+2) day and 30 (+/- 5) day observation
  number of deaths
Infection | based on 24-48 hour, 7 (-0/+2) day and 30 (+/- 5) day observation
  assessment of the wound left by the device implantation, considering any swelling of tissues around the device, fluctuation, redness, pain, excessive temperature, the outflow of any fluid from the pocket, CRP examination, WBC in the complete blood count

CONTACTS AND LOCATIONS:
Overall Officials: Przemysław Mitkowski, Prof. MD PhD, Principal Investigator — Medical University in Poznań
Locations (7):
- Poland (7):
  - I Cardiology Clinic, Medical University in Poznań, Poznan
  - Wolski Hospital, Cardiology Ward, Warsaw
  - Cardiology Clinic, Medical University of Warsaw, Warsaw
  - Clinical Department of Cardiology, the National Medical Institute of the Ministry of the Interior and Administration, Warsaw
  - I Clinic for Cardiac Arrhythmias National Institute of Cardiology Stefan Cardinal Wyszyński National Research Institute, Warsaw
  - Department of Cardiology / 1st Department of Cardiology and Angiology, Silesian Centre for Heart Diseases, Zabrze
  - Electrocardiology Clinic, Medical University, Lodz, Łódź Voivodeship

IPD SHARING:
Plan to Share IPD: No